CLINICAL TRIAL: NCT04181723
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Trofinetide for the Treatment of Girls and Women With Rett Syndrome
Brief Title: Study of Trofinetide for the Treatment of Girls and Women With Rett Syndrome (LAVENDER™)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-2566-003
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — trofinetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug - Trofinetide (Experimental): Trofinetide solution of 30-60 mL based on the subject's weight at Baseline, administered twice daily by mouth or gastrostomy tube (G-tube)
  Interventions: Drug: Trofinetide
- Placebo (Placebo Comparator): Trofinetide placebo solution of 30-60 mL based on the subject's weight at Baseline, administered twice daily by mouth or gastrostomy tube (G-tube)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Trofinetide — Trofinetide solution administered based on the subject's weight at Baseline, twice daily for 12 weeks
  Arms: Drug - Trofinetide
Other: Placebo — Trofinetide placebo solution administered based on the subject's weight at Baseline, twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
To investigate the efficacy of treatment with oral trofinetide versus placebo in females with Rett syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects 5 to 20 years of age, inclusive, at Screening
2. Body weight ≥12 kg at Screening
3. Can swallow the study medication provided as a liquid solution or can take it by gastrostomy tube
4. Has classic/typical Rett syndrome (RTT)
5. Has a documented disease-causing mutation in the MECP2 gene
6. Has a stable pattern of seizures, or has had no seizures, within 8 weeks of Screening
7. Subjects of childbearing potential must abstain from sexual activity for the duration of the study and for at least 30 days thereafter or must agree to use acceptable methods of contraception. Subject must not be pregnant or breastfeeding.
8. The subject's caregiver is English-speaking and has sufficient language skills to complete the caregiver assessments
9. Subject and caregiver(s) must reside at a location to which study drug can be delivered and have been at their present residence for at least 3 months prior to Screening

Exclusion Criteria:

1. Has been treated with insulin within 12 weeks of Baseline
2. Has current clinically significant cardiovascular, endocrine (such as hypo- or hyperthyroidism, Type 1 diabetes mellitus, or uncontrolled Type 2 diabetes mellitus), renal, hepatic, respiratory or gastrointestinal disease (such as celiac disease or inflammatory bowel disease) or has major surgery planned during the study
3. Has a history of, or current, cerebrovascular disease or brain trauma
4. Has significant, uncorrected visual or uncorrected hearing impairment
5. Has a history of, or current, malignancy
6. Has a known history or symptoms of long QT syndrome

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and condition do not meet all pre-specified entry criteria).

Ages: 5 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 187 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Translational Gemomics Research Institute (TGen), Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - UC Davis MIND Institute, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children Medical Services, Tampa, Florida
  - Emory Genetics Clinical Trial Center, Atlanta, Georgia
  - Rush University Children's Hospital, Chicago, Illinois
  - Kennedy Krieger Institute - Clinical Trials Unit, Baltimore, Maryland
  - Boston Children's Hospital Harvard Medical School, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center, Children's Hospital at Montefiore, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's, Seattle, Washington

REFERENCES:
- [Derived] Darwish M, Passarell J, Youakim JM, Bradley H, Bishop KM. Exposure-Response Efficacy Modeling to Support Trofinetide Dosing in Individuals with Rett Syndrome. Adv Ther. 2024 Apr;41(4):1462-1480. doi: 10.1007/s12325-024-02796-y. Epub 2024 Feb 16. PMID 38363467
- [Derived] Parent H, Ferranti A, Niswender C. Trofinetide: a pioneering treatment for Rett syndrome. Trends Pharmacol Sci. 2023 Oct;44(10):740-741. doi: 10.1016/j.tips.2023.06.008. Epub 2023 Jul 16. PMID 37460385
- [Derived] Neul JL, Percy AK, Benke TA, Berry-Kravis EM, Glaze DG, Marsh ED, Lin T, Stankovic S, Bishop KM, Youakim JM. Trofinetide for the treatment of Rett syndrome: a randomized phase 3 study. Nat Med. 2023 Jun;29(6):1468-1475. doi: 10.1038/s41591-023-02398-1. Epub 2023 Jun 8. PMID 37291210
- [Derived] Neul JL, Percy AK, Benke TA, Berry-Kravis EM, Glaze DG, Peters SU, Jones NE, Youakim JM. Design and outcome measures of LAVENDER, a phase 3 study of trofinetide for Rett syndrome. Contemp Clin Trials. 2022 Mar;114:106704. doi: 10.1016/j.cct.2022.106704. Epub 2022 Feb 8. PMID 35149233

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug - Trofinetide | Placebo
Started | 93 | 94
Completed | 70 | 85
Not Completed | 23 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug - Trofinetide | Placebo | Total
Number analyzed (Participants) | 93 | 94 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 85 | 89 | 174
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (4.69) | 10.9 (4.57) | 10.9 (4.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 94 | 187
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 17
  Not Hispanic or Latino | 86 | 84 | 170
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 82 | 90 | 172
  Black or African American | 1 | 1 | 2
  Asian | 5 | 1 | 6
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 93 | 94 | 187

OUTCOME MEASURES:

1. Primary Outcome: Rett Syndrome Behaviour Questionnaire (RSBQ) Total Score - Change From Baseline to Week 12
Description: The RSBQ is a 45-item caregiver-completed rating scale that includes 45 items, 39 of them grouped into 8 subscales, whose ratings reflect the severity and frequency of symptoms. Items are rated as 0 (not true), 1 (somewhat or sometimes true), or 2 (very true). The 8 subscales are general mood, breathing problems, hand behavior, face movements, body rocking/expressionless face, night-time behaviors, fear/anxiety, and walking/standing. Scores for item 31 are reversed in the calculation of the total score. The total score ranges from 0 to 90 and is calculated as the sum of the item scores. Higher scores mean worse behaviour.
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | -4.9 (0.94) | -1.7 (0.90)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.0175, Mixed-effects model for repeated measure; LSM difference = -3.1, 95% CI 2-sided [-5.7 to -0.6], Standard Error of Mean 1.30

2. Primary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at Week 12
Description: To rate how much the subject's illness has improved or worsened relative to a baseline state, a 7-point scale is used from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | 3.5 (0.07) | 3.8 (0.07)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.0030, Mixed-effects model for repeated measure; LSM difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.10

3. Secondary Outcome: Change From Baseline to Week 12 in Communication and Symbolic Behavior Scales Developmental Profile™ Infant-Toddler Checklist - Social Composite Score (CSBS-DP-IT Social)
Description: Standardized screening scale for assessing communication and pre-linguistic skills in young children 12-24 months and can be used with older children with developmental delay. The CSBS-DP includes a suite of three separate measures: The Infant-Toddler Checklist, a follow-up Caregiver Questionnaire and a Behavior Sample. In this study only the Infant-Toddler (CSBS-DP-IT) Checklist was used. The CSBS-DP-IT Checklist is a 24-item rating scale and each item is scored using a three-level rating of frequency: "not yet", "sometimes" and "often". The CSBS-DP-IT Social Composite score the range was 0 to 26 and a higher score represented a worse outcome. Three composite scores can be calculated: 1) Social Composite; 2) Speech Composite; 3) Symbolic Composite.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | -0.1 (0.26) | -1.1 (0.25)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.0064, Mixed-effects model for repeated measure; LSM difference = 1.0, 95% CI 2-sided [0.3 to 1.7], Standard Error of Mean 0.37

4. Secondary Outcome: Change From Baseline to Week 12 in Impact of Childhood Neurologic Disability Scale (ICND) Total Score
Description: The Impact of Childhood Neurologic Disability (ICND) scale evaluates the effect of four conditions or health problems on 11 aspects of a child's or family's life as "A lot", "Some", "A little", "Not at all", or "Does not apply". The four conditions or health problems are 1) inattentiveness, impulsivity, or mood, 2) ability to think and remember, 3) neurologic or physical limitations, and 4) epilepsy. The ICND score the range of 0 to 132 and a higher score represents a worse outcome.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | -6.5 (3.44) | -1.9 (3.14)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.3376, ANCOVA; LSM difference = -4.5, 95% CI 2-sided [-13.8 to 4.8], Standard Error of Mean 4.67

5. Secondary Outcome: Change From Baseline to Week 12 in Rett Syndrome Clinician Rating of Hand Function (RTT-HF)
Description: Clinical assessment of the subject's ability to use their hands for functional purposes (such as reaching for and grasping objects, self-feeding, or drawing). The assessment is made on an 8-point Likert scale (0-7) with 0 denoting normal functioning and 7 the most severe impairment.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | -0.1 (0.08) | 0.0 (0.07)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.3649, Mixed-effects model for repeated measure; LSM difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.11

6. Secondary Outcome: Change From Baseline to Week 12 in Rett Syndrome Clinician Rating of Ambulation and Gross Motor Skills (RTT-AMB)
Description: Clinical assessment of the subject's ability to sit, stand, and ambulate (e.g., walking, running, and climbing stairs). The assessment was made on an 8-point Likert scale (0 to 7), with 0 denoting normal functioning and 7 as the most severe impairment.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | -0.2 (0.07) | 0.0 (0.07)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.2114, Mixed-effects model for repeated measure; LSM difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.10

7. Secondary Outcome: Change From Baseline to Week 12 in Rett Syndrome Clinician Rating of Ability to Communicate Choices (RTT-COMC)
Description: Clinical assessment of the subject's ability to communicate their choices or preferences, which can include the use of nonverbal means such as eye contact or gestures. The assessment is made on an 8-point Likert scale (0-7) with 0 denoting normal functioning and 7 the most severe impairment.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | -0.4 (0.11) | 0.0 (0.10)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.0257, Mixed-effects model for repeated measure; LSM difference = -0.3, 95% CI 2-sided [-0.6 to 0.0], Standard Error of Mean 0.15

8. Secondary Outcome: Change From Baseline to Week 12 in Rett Syndrome Clinician Rating of Verbal Communication (RTT-VCOM)
Description: Clinical assessment of the subject's ability to communicate verbally (e.g. words and phrases). The assessment is made on an 8-point Likert scale (0-7) with 0 denoting normal functioning and 7 the most severe impairment.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | 0.0 (0.06) | 0.0 (0.06)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.9799, Mixed-effects model for repeated measure; LSM difference = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.08

9. Secondary Outcome: Change From Baseline to Week 12 in Clinical Global Impression-Severity (CGI-S)
Description: A 7 point scale that rates the severity of the subject's illness at the time of assessment, relative to the clinician's experience with subjects who have the same diagnosis. A subject is assessed on severity of illness at the time of rating: 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | 0.0 (0.03) | 0.0 (0.03)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.5304, Mixed-effects model for repeated measure; LSM difference = 0.0, 95% CI 2-sided [-0.1 to 0.1], Standard Error of Mean 0.05

10. Secondary Outcome: Change From Baseline to Week 12 in Rett Syndrome Caregiver Burden Inventory (RTT-CBI) Total Score (Items 1-24)
Description: The Rett Syndrome Caregiver Burden Inventory (RTT-CBI) scale is intended to directly address caregiver burden and indirectly assess the significance of treatment effects on function in the context of activities of daily living. Ratings are on a 5-point Likert scale including: 0-never; 1-rarely; 2-sometimes; 3-frequently and 4-nearly always. As in the original Caregiver Burden Inventory, the RTT-CBI has 24 negatively worded items (items 1 through 24) yielding a total score up to 96. The RTT-CBI the range is 0 to 96 and a higher score represents a worse outcome.
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | -1.1 (1.01) | -0.4 (0.96)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.5855, ANCOVA; LSM difference = -0.8, 95% CI 2-sided [-3.5 to 2.0], Standard Error of Mean 1.40

11. Secondary Outcome: Change From Baseline to Week 12 in Overall Quality of Life Rating of the Impact of Childhood Neurologic Disability Scale (ICND)
Description: The overall quality of life of the subject is also rated by responding to the following: "Please rate your child's overall 'Quality of Life' on the scale below. Choose the number which you feel is best and circle it." The choices range from 1 ("Poor") to 6 ("Excellent").
Time Frame: 12 Weeks Treatment Duration
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - Trofinetide | Placebo
Number analyzed (Participants) | 91 | 93
score on a scale | 0.2 (0.09) | 0.1 (0.09)
Statistical Analysis 1: Comparison: Drug - Trofinetide vs Placebo; Test type: Superiority; p = 0.2507, Mixed-effects model for repeated measure; LSM difference = 0.1, 95% CI 2-sided [-0.1 to 0.4], Standard Error of Mean 0.13

ADVERSE EVENTS:
Time Frame: Approximately 4 months
Arm/Group | Drug - Trofinetide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/94
Serious Adverse Events (participants affected / at risk) | 3/93 | 3/94
Other Adverse Events (participants affected / at risk) | 81/93 | 32/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug - Trofinetide (N=93) | Placebo (N=94)
Constipation (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug - Trofinetide (N=93) | Placebo (N=94)
Diarrhoea (Gastrointestinal disorders) | 75 | 18
Vomiting (Gastrointestinal disorders) | 25 | 9
Pyrexia (General disorders) | 8 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2
Seizure (Nervous system disorders) | 7 | 5
Irritability (Psychiatric disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT04181723/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT04181723/SAP_001.pdf